CLINICAL TRIAL: NCT02783157
Title: Transcutaneous Autonomic Modulation to Prevent Organ Injury After Thoracic Surgery
Brief Title: Transcutaneous Autonomic Modulation in Thoracic Surgery
Acronym: TON-POINTS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Pro00071148
Record Dates: First submitted 2016-04-13; First posted 2016-05-26 (Estimated); Last update posted 2020-04-06 (Actual); Status verified 2020-04

CONDITIONS: Atrial Fibrillation, Postoperative; Postoperative Complications; Inflammation
Keywords: Autonomic; Vagal nerve stimulation; Postoperative atrial fibrillation
MeSH Terms: conditions — Atrial Fibrillation; Postoperative Complications; Inflammation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcutaneous low-level vagal nerve stimulation (LLVNS) (Experimental): n=100 patients will be randomized to transcutaneous low-level vagal nerve stimulation (LLVNS), via a clip applied to the ear. Stimulation will be delivered throughout the procedure.
  Interventions: Device: Transcutaneous Low-Level Vagal Nerve Stimulation (LLVNS)
- Sham LLVNS (Sham Comparator): n=100 patients will be randomized to sham LLVNS, with the clip applied but no stimulation delivered.
  Interventions: Device: Sham LLVNS

INTERVENTIONS:
Device: Transcutaneous Low-Level Vagal Nerve Stimulation (LLVNS) — Low-level vagal nerve stimulation will be delivered via a clip applied to the ear throughout the surgical procedure. The voltage used will be individualized to each patient, based upon the voltage necessary to slow the sinus rate during testing.
  Arms: Transcutaneous low-level vagal nerve stimulation (LLVNS)
Device: Sham LLVNS — A clip will be applied to the ear, but no stimulation will be delivered throughout the procedure.
  Arms: Sham LLVNS

SUMMARY:
In this study, the investigators aim to determine whether non-invasive autonomic modulation decreases inflammation and complications after thoracic surgery. The investigators will test the hypothesis that low-level transcutaneous vagal nerve stimulation (LLVNS) during major thoracic surgery reduces inflammation and complications, particularly postoperative atrial fibrillation (POAF). This will be a prospective randomized pilot trial of 200 patients undergoing major thoracic surgery including lobectomy, bilobectomy, or pneumonectomy via either video-assisted thoracoscopic (VAT) or open thoracotomy. Patients will be randomized to receive ether a) LLVNS (n=100) or b) sham LLVNS (n=100) during their procedure. All patients will receive standardized anesthetic, surgical, and post-surgical care. The primary outcome in this study will be time to occurrence of in-hospital POAF, which will be compared between groups using Cox proportional hazards models. Secondary outcomes will be ICU and hospital length of stay, postoperative morbidity, postoperative mortality, and serologic markers of inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Major thoracic surgery (lobectomy, bilobectomy, or pneumonectomy via either video-assisted thoracoscopic (VAT) or open thoracotomy)

Exclusion Criteria:

* Patients >90 or <40 years of age
* Chronic atrial fibrillation
* Prior splenectomy
* Preoperative inotropic support
* Hepatic or renal failure
* Currently receiving vagal nerve stimulation therapy
* Taking centrally-acting cholinergic medications (tacrine, donepezil, rivastigmine)
* High-grade atrioventricular block (>2nd degree atrioventricular blockade)

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-05; Primary Completion 2020-02-21 (Actual); Study Completion 2020-02-21 (Actual)

PRIMARY OUTCOMES:
Incidence/Burden of Postoperative Atrial Fibrillation | Inpatient hospitalization approximately 3 to 7 days

SECONDARY OUTCOMES:
Postoperative morbidity | Inpatient hospitalization approximately 3 to 7 days, and one year after surgery
  The incidence of complications during the index hospitalization and one year after surgery
Postoperative mortality | Inpatient hospitalization approximately 3 to 7 days, and one year after surgery
  The incidence of complications during the index hospitalization and one year after surgery
Serologic Markers of Inflammation | Inpatient hospitalization approximately 3 to 7 days
  Cytokine levels, measured in pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: Joseph P Mathew, MD, MHS, MBA, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Stavrakis S, Humphrey MB, Scherlag BJ, Hu Y, Jackman WM, Nakagawa H, Lockwood D, Lazzara R, Po SS. Low-level transcutaneous electrical vagus nerve stimulation suppresses atrial fibrillation. J Am Coll Cardiol. 2015 Mar 10;65(9):867-75. doi: 10.1016/j.jacc.2014.12.026. PMID 25744003